CLINICAL TRIAL: NCT06038097
Title: Efficacy and Safety of Radiofrequency Pallidotomy in the Management of Dystonia - A Delayed Start Randomized Controlled Trial
Brief Title: Efficacy and Safety of Radiofrequency Pallidotomy in the Management of Dystonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC-465/03.08.2023
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Dystonia
Keywords: Dystonia; Segmental dystonia; Generalized dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention arm (Experimental): Radiofrequency Pallidotomy at earliest available date
  Interventions: Procedure: Radiofrequency Pallidotomy
- Delayed intervention arm (No Intervention): Radiofrequency pallidotomy offered at 12 weeks following agreeing to participate in the study

INTERVENTIONS:
Procedure: Radiofrequency Pallidotomy — Radiofrequency bilateral simultaneous pallidotomy
  Arms: Early intervention arm

SUMMARY:
Generalized dystonia is treated with pallidotomy. This is based on observational data which is significantly limited by publication bias and there are no RCTs. The case reports focus on successful outcomes and case series have an inherent selection bias. Bilateral pallidotomy has been used in our institute in a series of patients with generalized and segmental dystonia and have been seen to show good efficacy. However, the existing literature suggests that it is also associated with dysphagia and dysarthria in some cases and thus simultaneous bilateral pallidotomy is not preferred in several centres. However, our center routinely performs simultaneous bilateral pallidotomy.

The response rates and compliations of the procedure have not been systematically studied in RCT and we need to generate data on the efficacy and safety of Pallidotomy on generalized and segmental dystonia. This randomized controlled trial will fill the void in knowledge in this field.

DETAILED DESCRIPTION:
Deep brain stimulation surgery (DBS) has become the standard of care for the management of generalized dystonia It has been shown in Randomized controlled trials to be effective and safe.1-3 Since the last 30 years, DBS has been used to treat a variety of patients with dystonias, which are of varying etiologies. However, the DBS is an expensive system, needs hardware implantation and regular programming. It is associated with surgical implantation which may lead to complications such as infection of the hardware, leads and electrodes. Since it is expensive, it is out of reach for the majority of the patients who pay out of pocket. It leads to increased healthcare costs because of the initial expenses for the implant as well as regular follow ups for programming. The programming is currently labour intensive and needs long hours of observation with trial and error to find the optimum programming settings for the individual patient. This may need the patient to be admitted in the inpatient setting or multiple outpatient visits for the patient, which can lead to loss of working hours and burden on the healthcare system. Before the introduction of DBS by Benabid, functional neurosurgery with lesioning procedures such as pallidotomy, thalamotomy, subthalamotomy were used to manage movement disorders such as dystonia, tremors and Parkinson disease. However after the advent of DBS, these procedures have taken a backseat. Also there are no randomized trials for the safety and efficacy of lesioning procedures in dystonias. The current practice in various centers of the world is to do unilateral pallidotomy in most cases of dystonia. Simultaneous bilateral pallidotomy is not preferred by several practitioners due to the risk of bulbar symptoms which may be irreversible in certain cases. However, our experience in our Institute suggests good outcomes in patients with various forms of focal and generalized dystonias undergoing simultaneous bilateral pallidotomy using radiofrequency ablation. Similarly we have done pallidotomy for genetic dystonias such as NBIAs, Wilson's disease who had disabling dystonias or medically refractory status dystonicus.4 However, the long term efficacy and safety of these patients is not clear as there are no registries or long term follow up data. We need a well conducted Randomized controlled trial to systematically collect data on the efficacy and safety of the intervention to generate meaningful information for patients and clinicians to understand the risks and benefits of the procedures and offer relevant information for clinical decision making.

Problem statement Evidence based management requires robust data to make clinical decisions. This data is derived from studies which may be observational or interventional. In the evidence pyramid, meta-analysis of randomized controlled trials is considered to be of the highest quality of evidence.

Generalized dystonia is treated with pallidotomy. This is based on observational data which is significantly limited by publication bias and there are no RCTs. The case reports focus on successful outcomes and case series have an inherent selection bias. Bilateral pallidotomy has been used in our institute in a series of patients with generalized and segmental dystonia and have been seen to show good efficacy. However, the existing literature suggests that it is also associated with dysphagia and dysarthria in some cases and thus simultaneous bilateral pallidotomy is not preferred in several centres. However, our center routinely performs simultaneous bilateral pallidotomy.

The response rates and compliations of the procedure have not been systematically studied in RCT and we need to generate data on the efficacy and safety of Pallidotomy on generalized and segmental dystonia. This randomized controlled trial will fill the void in knowledge in this field.

Review of literature There are no randomized controlled trials to study the efficacy and safety of pallidotomy or thalamotomy in the management of dystonia. The case series and case reports regarding pallidotomy in dystonia describe a heterogenous population of patients who had undergone the procedure.5-10 Most of the case series have a bias towards reporting favourable outcomes. We found a meta-analysis of 100 patients who underwent bilateral procedures for dystonia.11 This meta-analysis described 33 studies with varying indications such as generalized dystonia, dystonic storm and focal dystonias. The majority of the patients had genetic causes of dystonia with DYT1 being the most common known genetic cause. Some studies reported a staged bilateral procedures while some simultaneous bilateral pallidotomy. The median time of follow up was 12 months with a range of 2-180 months. This meta-analysis revealed that 8% patients had transient adverse effects while 11% had permanent adverse effects. The commonest adverse effects that were permanent involved bulbar dysfunction with dysarthria anarthria or mutism. Most of the patients had a lasting beneficial effect while 19% patients had relapse of symptoms on prolonged follow up. The time to relapse of symptoms ranged from 3 weeks to 4.5 years. The predictors of response or relapse were not apparent from this meta-analysis. Moreover, why pallidotomy was preferred in contrast to DBS is not clear from the reports. Another case series describing 89 patients who underwent radiofrequency pallidotomy suggested unacceptable rates of complications with bilateral pallidotomy such as medically refractory parkinsonism, dysarthria and dysphagia.12 However these are retrospective review of data and the adverse effects may have been selectively reported in both unilateral and bilateral cases. In our center 10 children underwent bilateral simultaneous pallidotomy over a 7 year period and it was found that two patients had undergone the procedure for medically refractory status dystonicus and both of them had resolution of the status dystonicus. Two patients with generalized dystonia had recurrence of symptoms over a follow up of 4.5 years while three had a sustained improvement of more than 40% improvement in BFMDRS.4

ELIGIBILITY:
Inclusion Criteria:

1. Patients with generalized, segmental or focal dystonias who are being considered for simultaneous bilateral radiofrequency pallidotomy.
2. Of all ages and gender

Exclusion Criteria:

1. Those who deny consent
2. Pregnant ladies and women of childbearing potential without adequate contraception
3. Those who have undergone botulinum toxin injection in the last 12 weeks or those who are being planned for the same in the upcoming 12 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
BFM Dystonia disability scale | 6 weeks
  To compare the BFM Dystonia disability scale 6 weeks following bilateral simultaneous radiofrequency pallidotomy (early treatment arm) with the BFM Dystonia disability scale 6 weeks following acceptance of the procedure in those who were randomized to undergo the procedure atleast 12 weeks after accepting the the procedure (delayed treatment arm)
Adverse effects: New onset or worsening Dysphagia or dysarthria | 12 weeks
  To study the incidence of new onset or worsening dysphagia or dysarthria in patients with dystonia undergoing bilateral simultaneous pallidotomy

SECONDARY OUTCOMES:
20% improvement in BFM Dystonia disability scale | 6 weeks
  To compare the proportion of patients having atleast 20% improvement in BFM Dystonia disability scale from baseline to 6 weeks following bilateral simultaneous radiofrequency pallidotomy(early treatment arm) with the proportion of patients with similar improvement from baseline to 6 weeks following acceptance of procedure in those who undergo surgery atleast 12 weeks after accepting the procedure (delayed treatment arm)
20% improvement in BFM Dystonia movement scale | 6 weeks
  To compare the proportion of patients having atleast 20% improvement in BFM Dystonia movement scale from baseline to 6 weeks following bilateral simultaneous radiofrequency pallidotomy (early treatment arm) with the proportion of patients with similar improvement from baseline to 6 weeks following acceptance of procedure in those who undergo surgery atleast 3 months after accepting the procedure (delayed treatment arm)
Adverse effects | 12 weeks
  To study the proportion of patients in early and delayed treatment arm who develop adverse effects during the 12 weeks following surgery or agreeing for surgery respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Arunmozhimaran Elavarasi, MD DM, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be shared on approaching through proper channel through ethics committee AIIMS, New Delhi
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Will become available after the project is completed, will be available for 5 years atleast after completition of the trial
Access Criteria: De-identified patient data will be shared on approaching through proper channel through ethics committee AIIMS, New Delhi